CLINICAL TRIAL: NCT01448928
Title: Drug Use Investigation of Zevalin
Brief Title: Zevalin Post-marketing Surveillance in Japan
Acronym: ZEVALIN-DUI
Status: Completed | Type: Observational
Sponsor: Spectrum Pharmaceuticals, Inc (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 15042
Record Dates: First submitted 2011-08-17; First posted 2011-10-07 (Estimated); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Non-Hodgkin's Lymphoma (NHL)
Keywords: Zevalin; CD20+; Non-Hodgkin's Lymphoma; Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Mantle-Cell | interventions — ibritumomab tiuxetan

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: [90]Y-ibritumomab tiuxetan (Zevalin, BAY86-5128)

INTERVENTIONS:
Drug: [90]Y-ibritumomab tiuxetan (Zevalin, BAY86-5128) — Patients who have received Zevalin for relapsed or refractory, CD20+, low grade B-cell non-Hodgkin's lymphoma and Mantle cell lymphoma.

SUMMARY:
This study is a regulatory post marketing surveillance in Japan, and it is a local prospective and observational study of patients who have received Zevalin for relapsed or refractory, CD20+, low grade B-cell non-Hodgkin's lymphoma and Mantle cell lymphoma. The objective of this study is to assess safety and efficacy of using Zevalin in clinical practice. This study is also all case investigation of which the enrollment period is five years, and all patients who received Zevalin will be recruited and followed 13 weeks after the administration.

ELIGIBILITY:
Inclusion Criteria:

Patients who received Zevalin for relapsed or refractory:

* CD20+
* low grade B-cell non-Hodgkin's lymphoma
* Mantle cell lymphoma

Exclusion Criteria:

* Patients who are contraindicated based on the product label

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 400cases: This study is all case investigation of which the enrollment period is five years, and all patients who received Zevalin for relapsed or refractory, CD20+, low grade B-cell non-Hodgkin's lymphoma and Mantle cell lymphoma will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2008-09 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse drug reactions in subjects who received Zevalin | After In-111 Zevalin administration, up to 13 weeks
Incidence of serious adverse events, especially secondary malignant tumors, in subjects who received Zevalin | After In-111 Zevalin administration, up to 8 years

SECONDARY OUTCOMES:
Incidence of adverse drug reactions in subpopulation in a variety of baseline data [such as demographic data, medical history data, clinical staging] | After In-111 Zevalin administration, up to 13 weeks
Effectiveness evaluation assessment [complete remission rate, complete remission uncertain rate, partial remission rate, stable disease rate, progression disease rate] by investigator-determined overall best response | After In-111 Zevalin administration, up to 13 weeks
Effectiveness evaluation assessment [progression free survival] by investigator-determined overall best response | After In-111 Zevalin administration, up to 8 years
Change in hemoglobin from baseline | After In-111 Zevalin administration, up to 13 weeks
Change in neutrophil from baseline | After In-111 Zevalin administration, up to 13 weeks
Change in platelet from baseline | After In-111 Zevalin administration, up to 13 weeks
Change in leukocyte from baseline | After In-111 Zevalin administration, up to 13 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Multiple Locations, Japan